CLINICAL TRIAL: NCT06893315
Title: Photobiomodulation Therapy for Pain and Healing in Episiotomies and Grade 2 and 3 Perineal Lacerations After Vaginal Delivery: An Observational Study.
Brief Title: Photobiomodulation for Episiotomies and Perineal Lacerations After Vaginal Delivery.
Status: Active, not recruiting | Type: Observational
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, Professor M.D. Ph.D. Rebeca Boltes Cecatto, University of Nove de Julho
Other Study IDs: LUIRRUARO
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Perineal Lacerations; Delivery, Obstetric; Episiotomy Wound; Photobiomodulation Therapy; Pain
Keywords: Photobiomodulation; Low-level Laser Therapy; Wound healing; Episiotomy; Pain; Perineal Lacerations
MeSH Terms: conditions — Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient normal vaginal delivery postpartum patients: Inpatient postpartum patients during the puerperium who experienced grade 2 or 3 perineal laceration or underwent episiotomy during normal vaginal delivery who were treated during hospitalization with the standard hospital protocol for pain and local wound healing, and who were offered the use of PBM as an additional therapy by standard hospital protocol.
  Interventions: Radiation: Photobiomodulation Therapy; Other: Hospital Standard Protocol of treatment for pain and healing

INTERVENTIONS:
Radiation: Photobiomodulation Therapy — Photobiomodulation (PBM) is a non-invasive therapy that uses low-level light, typically from lasers or Light Emission Diodes (LEDs), to stimulate cellular function and promote healing. It works by delivering specific wavelengths of light to target tissues, which enhances mitochondrial activity and increases adenosine triphosphate (ATP) production. PBM is commonly used for pain relief, reducing inflammation, and accelerating tissue repair in conditions like muscle injuries, arthritis, and skin disorders.
Other: Hospital Standard Protocol of treatment for pain and healing — Medical team evaluations are conducted daily throughout the hospitalization period, and anti-inflammatory medications (ketoprofen ), analgesics (dipyrone), and, in cases where vulvar edema is observed, ice packs are prescribed. In addition to the standard treatment described, the health care team routinely offers patients the use of laser therapy (photobiomodulation) once a day during hospitalization. Patients who agree to the laser therapy receive both treatments.Patients who do not accept receiving PBM receive exactly only the same standard routine care described. These protocols are standardized at the hospital, and this observational study did not interfere with any care practices.

SUMMARY:
Episiotomies (EP) and perineal lacerations (PL) following vaginal delivery can lead to complications such as pain, edema, and infection. Currently, anti-inflammatory drugs, analgesics, baths, and ice packs are recommended for treatment. Photobiomodulation therapy (PBM) has emerged as a promising technology for pain management and scar healing in EP and PL. This is a cohort observational study conducted at the Maternal and Child University Hospital of the Universidade Estadual de Ponta Grossa, Paraná, Brazil. PBM adjuvant therapy is routinely applied at the bedside daily throughout the postpartum hospitalization. PBM is routinely offered to all postpartum patients during hospitalization. Patients may choose to accept or decline the use of analgesic PBM in addition to the standard therapeutic measures provided by the hospital (anti-inflammatory drugs, analgesics, baths, and ice packs). All patients who underwent EP or suffered grade 2 and 3 PL over six months are evaluated. We will analyze the data from patients who accepted the use of PBM and those who declined the use of PBM regarding the presence of pain, local healing of perineal lacerations, and episiotomies. The primary outcome is the daily pain assessment using the Numerical Pain Scale (NPS) before and after PBM (hospital standard). The secondary outcome is the evaluation of perineal healing using the REEDA scale. Initially, data distribution will be tested using the Kolmogorov-Smirnov test. Comparisons of NPS and REEDA scores between groups that received laser therapy and those that did not received will be performed using repeated-measures ANOVA, considering study covariates. Epidemiological and clinical data (age, sex, marital conditions, type and characteristics of labour (spontaneous or induced), newborn weight, presence of clinical complications during hospitalization ) collected directly in the patients' medical records to characterize the sample. All analyses will be conducted using SPSS 24.0 software, with a significance level of 95%.

DETAILED DESCRIPTION:
Episiotomies (EP) and perineal lacerations (PL) following vaginal delivery can lead to complications such as pain, edema, and infection. Currently, anti-inflammatory drugs, analgesics, baths, and ice packs are recommended for treatment. Photobiomodulation therapy (PBM) has emerged as a promising technology for pain management and scar healing in EP and PL. This is a cohort observational study conducted at the Maternal and Child University Hospital of the Universidade Estadual de Ponta Grossa, Paraná, Brazil. PBM therapy is routinely applied at the bedside daily throughout the postpartum hospitalization. It is standard practice at the hospital to offer adjuvant PBM in addition to the standard treatment (anti-inflammatory drugs, analgesics, baths, and ice packs). However, the use of PBM is optional for patients during hospitalization. The PBM parameters are: laser with a wavelength of 808 nm and a power of 100 mW applied at 5 points around the PL or EP for a total application time of 5 minutes. PBM is routinely offered to all postpartum patients during hospitalization. Patients may choose to accept or decline the use of analgesic PBM in addition to the standard therapeutic measures provided by the hospital (anti-inflammatory drugs, analgesics, baths, and ice packs). All patients who underwent EP or suffered grade 2 and 3 PL over six months period are evaluated. Since PBM is routinely offered to patients, after approval by the ethics committee, the principal investigator, monitored all included participants at the hospital and collected routine hospital data from medical records regarding the outcomes. We will analyze the medical record data related to the outcomes for statistical analysis. We will analyze the data from patients who accepted the use of PBM and those who declined the use of PBM regarding the presence of pain, local healing of perineal lacerations, and episiotomies. The outcomes will be analyzed by comparing the following participant subgroups: 1. participants who declined to receive PBM in addition to the hospital's standard treatment, and 2. participants who accepted to receive PBM in addition to the hospital's standard treatment. The primary outcome is the daily pain assessment using the Numerical Pain Scale (NPS) before and after PBM (hospital standard). The secondary outcome is the evaluation of perineal healing using the REEDA scale. Initially, data distribution will be tested using the Kolmogorov-Smirnov test. Comparisons of NPS and REEDA scores between groups that received laser therapy and those that did not will be performed using repeated-measures ANOVA, considering study covariates. All analyses will be conducted using SPSS 24.0 software, with a significance level of 95%. Epidemiological and clinical data (age, sex, marital conditions, type and characteristics of labour (spontaneous or induced), newborn weight, presence of clinical complications during hospitalization ) collected directly in the patients' medical records to characterize the sample and evaluate factors influencing the response to PBM regarding the assessed outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult women over 18 years of age;
* Parturients with a gestational age equal to or greater than 37 weeks;
* Patients who had a vaginal birth;
* Patients undergoing episiotomy or patients who presented grade 2 or 3 perineal laceration during childbirth.

Exclusion Criteria:

* Multiple pregnancy (twins);
* Presence of fetal malformation or death identified during prenatal care or at the time of hospitalization for delivery;
* Patients with serious complications such as severe puerperal hemorrhage or HELLP Syndrome during childbirth.
* Patients with grade 1 or 4 perineal lacerations.
* Presence of systemic diseases that alter the repair process.
* Withdrawal of the nformed Consent Form" (ICF) at the request of the patient or those responsible;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women in labor
Study Population: Patients undergoing episiotomy or patients who presented grade 2 or 3 perineal laceration during vaginal childbirth. The diagnosis of the degree of laceration is clinical and the obstetrician responsible for the patient's care treatment did so by exploring the injury and visualizing the injured structures within the hospital's care routine. Only those patients in whom the diagnosis of grade 2 or 3 perineal laceration made by the responsible care team and documented in the medical record were invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cutaneous pain | before and after each PBM session during the 3 days of hospitalization
  Perception of local cutaneous pain in the perineum, assessed daily by physiotherapists before and after each PBM session by Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Assessment of perineal lesion healing | Daily during hospitalization (3 days)
  Assessment of perineal lesion healing using the REEDA scale daily

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, PhD, Study Director — University of Nove de Julho
Locations (1):
- Hospital Universitário Materno-Infantil da Universidade Estadual de Ponta Grossa, Ponta Grossa, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The raw data without identification of these patients will be saved in an open access repository such as Mendeley Data or similar. The results of this study, whether favorable or not, will be published in impact journals.
Supporting Information: Study Protocol
Time Frame: after analysis of results
Access Criteria: The raw data without identification of these patients will be saved in an open access repository such as Mendeley Data or similar. The results of this study, whether favorable or not, will be published in impact journals.